CLINICAL TRIAL: NCT00174447
Title: Open Extension Study Evaluating The Long Term Efficacy , Safety And Tolerability Of Oral Ziprasidone In The Treatment Of Patients Who Have Successfully Completed The Previous Ziprasidone Study A1281031
Brief Title: Extension Study of Patients Successfully Treated by Ziprasidone in Study A1281031
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281060
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2009-11-17 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A1 (Experimental)
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — Dosage may subsequently be adjusted according to clinical status, only at each protocol visit and step by step between 40, 60 and 80 mg bid

SUMMARY:
Open label extension study of Ziprasidone, evaluation of safety of long term use of ziprasidone

ELIGIBILITY:
Inclusion Criteria:

* Patients who successfully completed study A1281031 (CGI score of 1 or 2 at final visit) or ZIP-NY-98035 and with QTc <= 500 msec.

Exclusion Criteria:

* All other patients who do not fit the inclusion criteria as stated above.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2001-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- France (13):
  - Pfizer Investigational Site, Avignon
  - Pfizer Investigational Site, DOLE Saint YLIE
  - Pfizer Investigational Site, Liévin
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Montfavet
  - Pfizer Investigational Site, Orvault
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Saint-Égrève
  - Pfizer Investigational Site, Saint-Rémy
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Toulon
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Versailles

REFERENCES:
- [Derived] Geier JL, Karayal ON, Lewis M, Camm JA, Keane M, Kremer CM, Kolluri S, Reynolds R, Eng S, Strom BL. Methodological challenges in the coding and adjudication of sudden deaths in a large simple trial with observational follow-up: the ziprasidone observational study of cardiac outcomes (ZODIAC). Pharmacoepidemiol Drug Saf. 2011 Nov;20(11):1192-8. doi: 10.1002/pds.2185. Epub 2011 Jul 27. PMID 21796719
- [Derived] Strom BL, Faich GA, Reynolds RF, Eng SM, D'Agostino RB, Ruskin JN, Kane JM. The Ziprasidone Observational Study of Cardiac Outcomes (ZODIAC): design and baseline subject characteristics. J Clin Psychiatry. 2008 Jan;69(1):114-21. doi: 10.4088/jcp.v69n0115. PMID 18312045
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281060&StudyName=Extension%20Study%20of%20Patients%20Successfully%20Treated%20by%20Ziprasidone%20in%20Study%20A1281031%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Ziprasidone: Ziprasidone maintenance dosing of 40 to 80 milligrams twice daily
Period: Overall Study
Arm/Group | Ziprasidone
Started | 43
Completed | 5
Not Completed | 38
Not completed — Adverse Event | 19
Not completed — Withdrawal by Subject | 15
Not completed — Protocol Violation | 1
Not completed — Lack of Efficacy | 1
Not completed — Administrative reason/Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ziprasidone
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Categorical Scores on Clinical Global Impression - Improvement (CGI-I)
Description: CGI-I consists of a 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale.
Time Frame: Baseline, 3 months, 6 months, 1 year, 3 years, 5 years, End of Study [LOCF]
Population: Intention to treat (ITT), all patients who received at least one dose of study medication and who have at least one post baseline efficacy evaluation. Imputation at Last Observation Carried Forward (LOCF).
Measure: Number; unit: participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 43
participants
  Baseline (n=43): very much improved | 13
  Baseline (n=43): much improved | 30
  3 months (n=35): very much improved | 10
  3 months (n=35): much improved | 20
  3 months (n=35): minimally improved | 2
  3 months (n=35): no change | 3
  6 months (n=34): very much improved | 11
  6 months (n=34): much improved | 18
  6 months (n=34): minimally improved | 2
  6 months (n=34): no change | 2
  6 months (n=34): minimally worsened | 1
  1 year (n=27): very much improved | 7
  1 year (n=27): much improved | 16
  1 year (n=27): minimally improved | 1
  1 year (n=27): no change | 3
  3 years (n=10): very much improved | 2
  3 years (n=10): much improved | 5
  3 years (n=10): no change | 2
  3 years (n=10): minimally worsened | 1
  5 years (n=7): very much improved | 2
  5 years (n=7): much improved | 4
  5 years (n=7): minimally improved | 1
  End of Study [LOCF] (n=43): very much improved | 5
  End of Study [LOCF] (n=43): much improved | 17
  End of Study [LOCF] (n=43): minimally improved | 5
  End of Study [LOCF] (n=43): no change | 6
  End of Study [LOCF] (n=43): minimally worsened | 4
  End of Study [LOCF] (n=43): much worsened | 6

2. Primary Outcome: Change From Baseline in CGI-I at End of Study (up to 5 Years)
Description: CGI-I consists of a 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Change from baseline is score at observation minus score at baseline.
Time Frame: Baseline, up to 5 years (End of Study [LOCF])
Population: ITT. LOCF.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 43
score on a scale | 1.4 (1.6)

3. Secondary Outcome: Number of Participants With Scores on Patient Preference Scale (PPS)
Description: Patient rated satisfaction scale with responses: Much better, I prefer this medication, Slightly better, About the same, Slightly worse, and Much worse, I much preferred my previous medication.
Time Frame: Baseline, up to 5 years (End of Study)
Population: ITT
Measure: Number; unit: participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 43
participants
  Baseline (n=43): much better | 28
  Baseline (n=43): slightly better | 13
  Baseline (n=43): about the same | 2
  End of study (n=28): much better | 4
  End of study (n=28): slightly better | 8
  End of study (n=28): about the same | 8
  End of study (n=28): slightly worse | 3
  End of study (n=28): much worse | 5

4. Secondary Outcome: Change From Baseline in Drug Attitude Inventory (DAI) at End of Study (up to 5 Years)
Description: DAI, a 10-item scale to assess how the attitude of schizophrenia patients toward their medications may affect compliance. Respondents indicate 'true' or 'false' for each item. An overall calculated score ranges from -10 to 10, where a positive score indicated a positive subjective response (compliant), whilst a negative score indicated non-compliance. Change: score at observation minus score at baseline.
Time Frame: Baseline, up to 5 years (End of Study)
Population: ITT. n= number of participants with analyzable data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 24
score on a scale | -3.3 (4.6)

5. Primary Outcome: Number of Participants With Categorical Scores on Clinical Global Impression of Severity (CGI-S)
Description: CGI-S Scale: standardized assessment tool to rate severity of subject's illness; assessed investigator's impression of subject's current illness state. Score: 1 (normal - not ill at all) to 7 (among the most extremely ill patients).
Time Frame: Baseline, 3 months, 6 months, 1 year, 3 years, 5 years, End of Study [LOCF]
Population: ITT. LOCF.
Measure: Number; unit: participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 43
participants
  Baseline (n=43): normal, not ill at all | 4
  Baseline (n=43): borderline | 20
  Baseline (n=43): mildly ill | 14
  Baseline (n=43): moderately ill | 4
  Baseline (n=43): markedly ill | 1
  3 months (n=35): normal, not ill at all | 6
  3 months (n=35): borderline | 13
  3 months (n=35): mildly ill | 10
  3 months (n=35): moderately ill | 6
  6 months (n=34): normal, not ill at all | 8
  6 months (n=34): borderline | 10
  6 months (n=34): mildly ill | 11
  6 months (n=34): moderately ill | 5
  1 year (n=27): normal, not ill at all | 6
  1 year (n=27): borderline | 10
  1 year (n=27): mildly ill | 9
  1 year (n=27): moderately ill | 2
  3 years (n=10): normal, not ill at all | 1
  3 years (n=10): borderline | 5
  3 years (n=10): mildly ill | 2
  3 years (n=10): moderately ill | 2
  5 years (n=7): normal, not ill at all | 1
  5 years (n=7): borderline | 4
  5 years (n=7): mildly ill | 2
  End of Study [LOCF] (n=43): normal, not ill at all | 4
  End of Study [LOCF] (n=43): borderline | 9
  End of Study [LOCF] (n=43): mildly ill | 9
  End of Study [LOCF] (n=43): moderately ill | 10
  End of Study [LOCF] (n=43):markedly ill | 8
  End of Study [LOCF] (n=43): severely ill | 3

6. Primary Outcome: Change From Baseline in CGI-S at End of Study (up to 5 Years)
Description: CGI-S Scale: standardized assessment tool to rate severity of subject's illness; assesses investigator's impression of subject's current illness state. Score: 1 (normal - not ill at all) to 7 (among the most extremely ill). Change: score at observation minus score at baseline.
Time Frame: Baseline, up to 5 years (End of Study [LOCF])
Population: ITT. LOCF.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 43
score on a scale | 0.9 (1.5)

ADVERSE EVENTS:
Arm/Group | Ziprasidone
Serious Adverse Events (participants affected / at risk) | 13/43
Other Adverse Events (participants affected / at risk) | 36/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=43)
Schizophrenia (Psychiatric disorders) | 4
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Drug abuse (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Schizoaffective disorder (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 2
Faecal incontinence (Gastrointestinal disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Memory impairment (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=43)
Anxiety (Psychiatric disorders) | 10
Schizophrenia (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 7
Depression (Psychiatric disorders) | 5
Depressed mood (Psychiatric disorders) | 5
Panic attack (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 2
Hallucination (Psychiatric disorders) | 2
Schizoaffective disorder (Psychiatric disorders) | 1
Abulia (Psychiatric disorders) | 1
Alcoholism (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 1
Libido increased (Psychiatric disorders) | 1
Middle insomnia (Psychiatric disorders) | 1
Psychomotor retardation (Psychiatric disorders) | 1
Reactive psychosis (Psychiatric disorders) | 1
Stress (Psychiatric disorders) | 1
Headache (Nervous system disorders) | 4
Extrapyramidal disorder (Nervous system disorders) | 2
Parkinsonism (Nervous system disorders) | 2
Sensory disturbance (Nervous system disorders) | 2
Akathisia (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Weight decreased (Investigations) | 5
Weight increased (Investigations) | 4
Influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Tongue disorder (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hypotension (Vascular disorders) | 4
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Drug dispensing error (Injury, poisoning and procedural complications) | 3
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 1
Asthenia (General disorders) | 3
Chest discomfort (General disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Deafness unilateral (Ear and labyrinth disorders) | 1
Myopia (Eye disorders) | 1
Visual disturbance (Eye disorders) | 1
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Breast cyst (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Tachycardia (Cardiac disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Langerhans' cell granulomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.